CLINICAL TRIAL: NCT02868931
Title: Evaluation of a Newly Developed Treatment and Education Program (INPUT) for Diabetic Patients Performing an Insulin Pump Therapy
Brief Title: Evaluation of a Diabetes Treatment and Education Program for Insulin Pump Therapy (INPUT)
Acronym: INPUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norbert Hermanns (Other)
Collaborators: Berlin-Chemie (Unknown)
Responsible Party: Sponsor-Investigator, Norbert Hermanns, CEO, Forschungsinstitut der Diabetes Akademie Mergentheim
Organization: Forschungsinstitut der Diabetes Akademie Mergentheim (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NH012016
Record Dates: First submitted 2016-04-20; First posted 2016-08-16 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus
Keywords: self-management; empowerment; treatment and education program; insulin pump; diabetes education
MeSH Terms: conditions — Diabetes Mellitus; Empowerment | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- INPUT (Experimental): INPUT consists of 12 lessons comprising all relevant information in order to treat diabetes with an insulin pump. Patients learn to effectively use the different features of their pump in order to improve not only glycemic control but also to improve the implementation of pump therapy in daily life. Psychological and motivational aspects of living with diabetes and living with an insulin pump are addressed as well.
  Interventions: Behavioral: INPUT
- Waiting list (No Intervention): Patients are randomly assigned to the waiting list. After completion of the 6-month follow-up, these patients will also receive training with INPUT.

INTERVENTIONS:
Behavioral: INPUT — Treatment and education program based on the self-management theory of behavioral medicine.
  The program is delivered by certified and specially trained diabetes educators.
  Other Names: treatment and education program for INsulin PUmp Therapy
  Arms: INPUT

SUMMARY:
This study is a randomized, controlled, prospective trial with a 6-month follow-up. A newly developed treatment and education programme for diabetic patients with an insulin pump therapy (INPUT) will be tested compared to a waiting group. Primary outcome variable is the difference in glycemic control between baseline and the 6-month follow-up. Secondary outcome variables are: severe hypoglycaemia, diabetes-related distress, depressive symptoms, health-related quality of life, diabetes empowerment, self-care behavior, hypoglycemia awareness, and attitudes towards insulin pump therapy.

DETAILED DESCRIPTION:
INPUT is a self-management-based treatment and education program for diabetic patients with an insulin pump (CSII). It is designed to empower patients to adequately perform their therapy in daily life and to integrate their diabetes and their insulin pump into their lifes in order to enhance quality of life.

INPUT ist tested in an randomized controlled trial (RCT) with a waiting-list control group since no certified and effective treatment and education program for CSII exists.

This study is a multi-center study. Study centers are specialized diabetes practices throughout Germany. Patients will be approached by their respective practice and informed about the study. Study measurements as well as the conduct of INPUT will take place at the respective practice.

Baseline measurement will take place 2 weeks prior to the beginning of INPUT. After completion of baseline measurement, all patients from one study center will be randomized centrally by the Research Institute of the Diabetes Academy Mergentheim (FIDAM). 2 weeks and 6 months after the completion of INPUT, follow-up measurements will be conducted at the respective study center.

HbA1c as a marker of glycemic control will be analyzed in a central laboratory. Secondary outcome measures will be assessed via psychometrically tested questionnaires, Case Reports Forms, or patient files.

ELIGIBILITY:
Inclusion Criteria:

* Existing insulin pump therapy
* Prior participation in a structured diabetes education program
* HbA1c ≥ 7,5% but ≤ 13%
* Ability to understand, speak and write German language
* informed consent (if necessary, informed consent of the parents)

Exclusion Criteria:

* Diabetes duration < 1 year
* severe organic disease preventing a regular participation in the training course
* pregnancy
* severe cognitive impairment
* current treatment of psychiatric disorder
* renal disease requiring dialysis

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Changes in Glycemic Control Measured by A1c | 6 months
  Difference between baseline A1c and A1c at the 6-month follow-up

SECONDARY OUTCOMES:
Hypoglycaemia Awareness | 6 months
  The hypoglycemia awareness questionnaire provides a score indicating the severity of hypoglycaemia unawareness. This scale ranges from 0 (maximum hypoglycaemia awareness) to 7 (minimum hypoglycaemia awareness), where a score of 4 suggests reduced hypoglycaemia awareness.
Diabetes Empowerment | 6 months
  Empowerment is measured by a German version of the Diabetes Empowerment Scale, a measure of diabetes-related psychosocial self-efficacy.
Satisfaction with current treatment | 6 months
  Satisfaction with current treatment is assessed via a 10-item scale. The total score ranges from 10 to 60 with lower scores indicating higher satisfaction.
Diabetes Self-Management | 6 months
  The Diabetes Self-Management Questionnaire is a self-report measure of patients' self-care. The level of self-care is assessed via Likert scales.
Diabetes Distress | 6 months
  The Diabetes Distress Scale (DDS) assesses diabetes-related stressors due to living and treating diabetes. Different aspects of distress are covered: emotional burden, physician-related, regimen-related, diabetes-related interpersonal
Problem Areas in Diabetes | 6 months
  The Problem Areas in Diabetes Scale (PAID) assesses the psychosocial adaptation to the burden of living with and treating diabetes.
Health-related Quality of Life | 6 months
  Health-related quality of life focuses on the health-specific aspects of quality of life and dealing with a chronic condition such as diabetes
Depressive symptoms | 6 months
  The presence and extent of typical depressive symptoms are assessed via self-report
Attitudes towards insulin pump therapy | 6 months
  Specific attitudes towards different aspects of insulin pump therapy are assessed via Likert scales. The questionnaire consists of 6 subscales that can be placed within 4 dimensions: (I) Expectations on insulin pump therapy (subscale: achieving better glycaemic control) (II) Perceived advantages of an insulin pump (subscale: gaining more flexibility) (III) Ease of use (subscales: design + functionality) (IV) Psychosocial effects and barriers (subscales: technological dependence + impaired body image)
Severe hypoglycaemia | 6 months
  The incidence of severe hypoglycaemia in the past six months is assessed via Case Report Forms. Severe hypoglycaemia is defined as requiring third party assistance or medical intervention for treating hypoglycaemia.

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Hermanns, PhD, Principal Investigator — Forschungsinstitut der Diabetes Akademie Mergentheim (FIDAM GmbH)
Locations (1):
- Diabetologische Schwerpunktpraxis Neuss, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ehrmann D, Kulzer B, Schipfer M, Lippmann-Grob B, Haak T, Hermanns N. Efficacy of an Education Program for People With Diabetes and Insulin Pump Treatment (INPUT): Results From a Randomized Controlled Trial. Diabetes Care. 2018 Dec;41(12):2453-2462. doi: 10.2337/dc18-0917. Epub 2018 Oct 10. PMID 30305343